CLINICAL TRIAL: NCT02569437
Title: The Role of Doxycycline in Management of Moderate to Severe Chronic Rhinosinusitis With Nasal Polyps
Brief Title: Doxycycline in Treating Patients With Chronic Rhinosinusitis With Nasal Polyps
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A high percentage of patients were dropping out of the study and were not able to complete the protocol.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Benjamin D Malkin, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 14-0462
Record Dates: First submitted 2015-10-05; First posted 2015-10-06 (Estimated); Results first posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-12

CONDITIONS: Polyp of Nasal Sinus
Keywords: doxycycline; oral methylprednisone; sinusitis with nasal polyps
MeSH Terms: interventions — Doxycycline; Methylprednisolone; Fluticasone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Doxycycline (Experimental): Doxycycline plus oral methylprednisolone and nasal saline sprays
  Interventions: Drug: Doxycycline; Drug: methylprednisolone; Drug: nasal saline spray; Drug: Flonase
- Sugar pill (Placebo Comparator): placebo pill plus oral methylprednisolone for three weeks. After this, maintenance therapy which includes nasal saline sprays and daily nasal steroid sprays.
  Interventions: Drug: methylprednisolone; Drug: Flonase; Drug: sugar pill

INTERVENTIONS:
Drug: Doxycycline — Doxycycline (200 mg PO X 1 dose on Day 1, then 100 mg PO daily) for Day 2-20
  Arms: Doxycycline
Drug: methylprednisolone — oral methylprednisolone: 32 mg x 5 days, 16 mg x 5 days, 8 mg x 10 days
Drug: nasal saline spray — nasal saline sprays: 2 sprays each nostril three times a day
  Arms: Doxycycline
Drug: Flonase — daily nasal steroid sprays (Flonase, 2 sprays each nostril daily).
  Other Names: nasal steroid spray
Drug: sugar pill — placebo pill to match doxycycline
  Other Names: placebo
  Arms: Sugar pill

SUMMARY:
The Department of Otolaryngology at Mount Sinai is looking for adults with sinus disease with polyps, otherwise called chronic rhinosinusitis with nasal polyps (CRSwNP). Patients may be eligible to enroll in a study offering a cutting-edge therapy to help reduce symptoms and avoid surgery. The treatment combines an antibiotic (doxycycline) with oral steroids. Oral steroids are the mainstay of medical management for patients with CRSwNP. However, recent studies have shown that doxycycline helps improve symptoms as well by reducing inflammation and killing common bacteria that can cause symptoms. This study is the first to evaluate this combination regimen.

DETAILED DESCRIPTION:
An eligible patient may be treated with either doxycycline and oral steroids OR placebo (sugar pill) and oral steroids for three weeks. Volunteers will participate in the study for to 12 weeks, and will have 4 research visits of 1 hour duration. At each study visit, the patient will under go an endoscopic evaluation and asked to complete a questionnaire describing symptoms. There is no additional cost to be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Nasal polyps on nasal endoscopy.
* The patient has moderate to severe disease, defined by moderate to severe subjective symptoms (a score greater than 3 on a 10-cm VAS).
* The patient is at least 18 years old.
* The patient is able to understand and give informed consent.
* The patient has clinically diagnosed chronic rhinosinusitis with nasal polyps according to the AAO-HNS diagnostic criteria: At least 2 of the following symptoms/signs:

  * Mucopurulent drainage (anterior, posterior, or both)
  * Nasal obstruction (congestion)
  * Facial pain-pressure-fullness
  * Decreased sense of smell
  * and symptoms lasting 12 weeks or longer.

Exclusion Criteria:

* The patient has a history of treatment with oral corticosteroids in the past 4 weeks. ,
* The patient has cystic fibrosis.
* The patient has primary ciliary dyskinesia.
* The patient has diabetes.
* The patient has had sinus surgery in the past 3 months.
* The patient has an allergy to doxycycline or related tetracyclines or glucocorticoids.
* The patient is a minor.
* The patient is a prisoner.
* The patient has a psychiatric illness or developmental delay, which would interfere with understanding of the study and provision of informed consent.
* The patient is a breastfeeding mother. The effects of the drugs used in this study (doxycycline) on breast milk are unknown and thus, these patients will be excluded from the study
* The patient has a history of HIV or other known cause of immunosuppression, or is actively taking immunosuppressive medications due to organ transplantation, rheumatoid disease, or other medical conditions.
* The patient is on penicillin; antacids containing aluminum, calcium, magnesium, or iron; bismuth subsalicylate; barbiturates; carbamazepine; and phenytoin; as well as tetracycline and Penthane.
* Pregnancy. Doxycycline, a tetracycline, is a known teratogen. For this reason women of child-bearing potential are suggested to take a form of contraception for the duration that they are taking doxycycline., Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Pregnancy Testing. Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) prior to the first dose of drug. No further pregnancy tests are required since after this visit the patient will no longer be taking tetracycline after 3 weeks.

Women of childbearing potential are defined as follows:

* Patients with regular menses
* Patients with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
* Women who have had a tubal ligation

Women are considered not to be of childbearing potential for the following reasons:

* The patient has undergone hysterectomy and/or bilateral oophorectomy.
* The patient is post-menopausal defined by amenorrhea for at least 1 year in a woman > 45 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-09; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Malkin, MD, Principal Investigator — Icahns School of Medicine at Mount Sinai; Satish Govindaraj, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from September 2014 to April 2016 at the Mount Sinai Department of Otolaryngology-Head & Neck Surgery rhinology practice.
Period: Overall Study
Arm/Group | Doxycycline | Sugar Pill
Started | 24 | 25
Completed | 12 | 11
Not Completed | 12 | 14
Not completed — Lost to Follow-up | 12 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxycycline | Sugar Pill | Total
Number analyzed (Participants) | 24 | 25 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (13.8) | 44.1 (12.2) | 47.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 14 | 12 | 26
Number of Participants with Prior Endoscopic Sinus Surgery (ESS) [Count of Participants; unit: Participants] | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Sino-nasal Outcome Test (SNOT 22)
Description: a validated 22 item quality of life questionnaire for patients with chronic rhinosinusitis. Range of 0 to 110, higher scores indicate worse outcome
Time Frame: Baseline and 12 weeks
Population: An additional 7 patients in the treatment group and 10 patients in the placebo group completed SNOT-22 scores via phone calls, even after study withdrawal.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Doxycycline | Sugar Pill
Number analyzed (Participants) | 24 | 25
units on a scale
  Baseline | 55.2 (24.3) | 54.4 (20.8)
  12 weeks: number analyzed (Participants) | 19 | 21
  12 weeks | 43.7 (6.2) | 49.8 (5.8)

2. Secondary Outcome: Endoscopic Nasal Polyp Score
Description: 0- Absence of nasal polyps
  1. Polyps confined to the middle meatus and not beyond the inferior border of the middle turbinate
  2. Polyps reaching below the lower border of the middle turbinate
  3. Large polyps extending to the lower border of the inferior turbinate or medial to the middle turbinate
  4. Large polyps extending to the lower border of the inferior turbinate or medial to the middle turbinate Nasal polyp scores. The score is determined for each nostril, and the two scores added for a total nasal polyp score. Range of 0 to 8, graded on a size system from 0 to 4 and summed from the right and left nostrils.
Time Frame: Baseline and 12 weeks
Population: There were 12 subject withdrawals in the treatment group and 14 in the placebo group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Doxycycline | Sugar Pill
Number analyzed (Participants) | 24 | 25
units on a scale
  Baseline | 6.0 (1.8) | 6.5 (1.3)
  12 weeks: number analyzed (Participants) | 12 | 11
  12 weeks | 4.3 (0.5) | 4.9 (0.5)

3. Secondary Outcome: Middle Meatus Culture
Description: Culture swab for the presence or absence of microbial growth
Time Frame: Baseline and 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Doxycycline | Sugar Pill
Number analyzed (Participants) | 24 | 25
Participants
  Culture growth at initial visit and 12 week visit | 5 | 2
  Culture growth initial visit, none at 12 weeks | 1 | 2
  No growth initial visit, but growth at 12 weeks | 2 | 1

4. Secondary Outcome: Subjective Symptom Composite Scoring
Description: A subjective symptom score will be extracted from the patient's score (on a scale of 0-5, where 0 defines no problems with the given symptom and 5 defines maximal problems ) on the SNOT-22 for each fo the following symptoms: "blockage/congestion," "runny nose," "post-nasal discharge," "facial pain/pressure," and "sense of taste/smell." Range of 0 to 25, with higher score reflecting worse symptoms.
Time Frame: Baseline and 12 weeks
Population: There were 12 subject withdrawals in the treatment group and 14 in the placebo group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Doxycycline | Sugar Pill
Number analyzed (Participants) | 24 | 25
units on a scale
  Baseline | 16.3 (5.2) | 17.1 (4.4)
  12 weeks: number analyzed (Participants) | 12 | 11
  12 weeks | 11.9 (1.5) | 13.6 (1.4)

5. Secondary Outcome: Visual Analog Scale
Description: The visual analog scale for overall symptoms will be used to define disease severity. Range of 0 to 10. As per the European Position Paper 2012, mild, moderate, and severe disease will be defined as 0 to and including 3, > 3 to and including 7, and > 7 to and including 10, respectively.
Time Frame: Baseline and 12 weeks
Population: There were 12 subject withdrawals in the treatment group and 14 in the placebo group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Doxycycline | Sugar Pill
Number analyzed (Participants) | 24 | 25
units on a scale
  Baseline | 8.4 (1.5) | 8.1 (1.3)
  12 weeks: number analyzed (Participants) | 12 | 11
  12 weeks | 5.2 (0.7) | 4.5 (0.7)

ADVERSE EVENTS:
Arm/Group | Doxycycline | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/25
Other Adverse Events (participants affected / at risk) | 0/24 | 0/25

LIMITATIONS AND CAVEATS:
Power not adequate and study is at risk for a Type II error - study was ended prior to complete sample size accrual. Study recruited high percentage of severe disease patients, thus did not accurately represent moderate disease patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes